CLINICAL TRIAL: NCT02210520
Title: Effect of Laser and Ultrasound in Pain and Disability in Women With Chronic Non-specific Low Back Pain: Randomized Double-blinded Controled Trial
Brief Title: Effect of Ultrasound and Laser in Chronic Low Back Pain: Randomized Double-blinded Controled Trial
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Ana Paula Fernandes A. Rubira, Master, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: São Lucas College
Record Dates: First submitted 2014-07-11; First posted 2014-08-06 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Lasers

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- laser (Experimental): 3 J/cm², 2 minutes in 6 points around the back spine
  Interventions: Device: pulsatile ultrasound; Device: continuous ultrasound
- pulsatile ultrasound (Experimental): 1 W/cm², 2 minutes in 6 points around the back spine
  Interventions: Device: continuous ultrasound; Device: laser
- continuous ultrasound (Experimental): 1 W/cm², 2 minutes in 6 points around the back spine, three times in the week, during 10 sessions per four weeks.
  Interventions: Device: pulsatile ultrasound; Device: laser
- control (No Intervention): no treatment.

INTERVENTIONS:
Device: pulsatile ultrasound — 1 W/cm², 2 minutes in 6 points around the back spine, three times in the week, during 10 sessions per four weeks.
  Arms: continuous ultrasound; laser
Device: continuous ultrasound — 1 W/cm², 2 minutes in 6 points around the back spine, three times in the week, during 10 sessions per four weeks.
  Arms: laser; pulsatile ultrasound
Device: laser — 1 W/cm², 2 minutes in 6 points around the back spine
  Arms: continuous ultrasound; pulsatile ultrasound

SUMMARY:
The low level laser therapy has a better effect in decrease the pain than ultrasound therapeutic.

DETAILED DESCRIPTION:
The laser will be applied with the dosimetry 3 J/cm², 2 minutes in 6 points around the back spine, during 4 weeks. Before the women will be evaluate again.

ELIGIBILITY:
Inclusion Criteria:

* chronic low back pain
* 3,0 - 7,0 in the visual analogic scale

Exclusion Criteria:

* no use of medications
* no other treatment
* without fractures, pregnancy, psychiatric or neurologic disorders, diabetes, amputations
* with diagnostic of low back pain

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 4 weeks
  Visual Analog Scale

SECONDARY OUTCOMES:
Pain quality | 4 weeks
  McGill questionaire
Disability | 4 Weeks
  Roland Morris Questionaire

CONTACTS AND LOCATIONS:
Overall Officials: Ana Paula A Rubira, master, Principal Investigator — São Paulo University
Locations (1):
- São Lucas College, Porto Velho, Rondõnia, Brazil